CLINICAL TRIAL: NCT03317600
Title: Postamputation Pain: Peripheral Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Nerveblock2017
Record Dates: First submitted 2017-10-13; First posted 2017-10-23 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Neuropathic Pain; Amputation, Traumatic; Nerve Block; Phantom Limb Pain; Stump Pain
MeSH Terms: conditions — Neuralgia; Amputation, Traumatic; Phantom Limb

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine block (Active Comparator)
  Interventions: Device: Lidocaine
- Isotonic saline block (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Lidocaine — Intervention is a nerve block with Lidocaine 2% with Adrenaline.
  Arms: Lidocaine block
Drug: Placebo — Intervention is a "placebo" nerve block with isotonic saline
  Arms: Isotonic saline block

SUMMARY:
Stump and phantom pain after amputation are common, but the responsible mechanisms are still not clarified. It has been suggested that phantom limb pain can be reduced by regional anaesthesia and in several recent studies, pain was reduced following intrathecal and intraforaminal blocks. In this study, the investigators want to investigate if spontaneous and evoked pain in amputees will be relieved by regional nerve blocks involving the damaged nerves.

ELIGIBILITY:
Inclusion Criteria:

* Amputees with chronic amputation pain (stump or phantom pain) 3 or above on NRS (numerical ratio scale).

Exclusion Criteria:

* Severe somatic or psychiatric diseases
* Other peripheral neuropathy
* Lack of ability to cooperate to the clinical examination
* Allergy to Lidocaine or similar analgetics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Reduction in spontaneous pain on a Numeric Rating Scale (NRS: 0-10, 0 = no pain, 10 = worst possible pain) | From 0 minutes until 120 minutes after injection
  The patient will be asked about spontaneous pain, including stump and phantom pain on a Numerical Rating Scale (NRS: 0-10, 0 = no pain, 10 = worst pain).

SECONDARY OUTCOMES:
Reduction in evoked pain on a Numerical Rating Scale (NRS: 0-10, 0 = no pain, 10 = worst possible pain). | From 0 minutes until 120 minutes after injection
  The patient will be asked about evoked pain on a Numerical Rating Scale (NRS: 0-10, 0 = no pain, 10 = worst pain). Evoked pain is triggered by a SOMEDIC brush, thermo rolls (20 degrees Celcius and 40 degrees Celcius) and pinprick with a von Frey filament (60 g).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark